CLINICAL TRIAL: NCT05441358
Title: Assessment of Platelet Function in Patients Undergoing Open Heart Surgery
Acronym: Saturn
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: LifeBridge Health (Other)
Collaborators: Sinai Center for Thrombosis Research and Drug Development (Unknown); Accriva Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: 1813901
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Coronary Artery Bypass Grafting; Open Heart Surgery; Aortic Surgery or Redo Surgery; On-pump Double or Triple Valve Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing open heart surgery: Subjects scheduled for elective cardiothoracic surgery requiring a sternotomy.
  * Coronary artery bypass grafting (CABG)
  * Combined CABG and valve surgery
  * On-pump double or triple valve procedures
  * Aortic surgery or redo surgery
  * Off pump CABG as part of a hybrid revascularization approach
  Interventions: Procedure: Open Heart Surgery

INTERVENTIONS:
Procedure: Open Heart Surgery — Blood collection at 4 timepoints (prior to anesthesia induction, immediately post-protamine, 1-2 hours post protamine, and up to 48 hours post-surgical completion) to assess platelet function.
  Other Names: CABG; Open Heart Valve Replacement

SUMMARY:
The purpose of this external evaluation is to assess the system functionality and analytical performance of the Saturn Investigational Instrument (next generation VerifyNow instrument) and associated cartridge currently under development.

A single test cartridge with multiple assays will be compared with Light Transmittance Aggregometry (LTA) within a clinical setting using blood samples. Analytical performance will be compared between these assays. The outcome of this evaluation will be used to demonstrate baseline performance and support the design and development of the Saturn analyzer and optimization of the associated algorithm.

DETAILED DESCRIPTION:
This protocol applies to the evaluation of the Saturn Investigational Instrument and cartridge. LTA will serve as the reference analyzer for this study. The evaluation will be conducted at Sinai Hospital ( Baltimore, Maryland).

The Sponsor has determined that this investigation is classified as a non-significant risk study. While there are risks associated with the cardiac procedure, there is minimal additional risk associated with having blood specimen collection during the standard of care operation.

Risks to the operator include potential exposure to blood-borne pathogens if a patient's blood specimen is infected. The risk is mitigated by only allowing trained personnel to participate in the study.

Results obtained from the investigational device shall not be used for any clinical assessments, decisions, or treatments for any subjects enrolled in the study, or any patients not enrolled in the study. No study-specific test results shall be provided to the subject. Study-specific test results will only be accessible by personnel duly trained to the study protocol and authorized for use of the study analyzers and/or study-specific data capture systems.

Project Saturn is the next generation VerifyNow System. The System includes an analyzer, single-use test cartridges, and associated quality controls. Project Saturn will be developed and commercialized in two phases. Phase 1 includes a modern analyzer which will perform the current, on-market VerifyNow Tests: PRUTest and Aspirin Test. Phase 2 will utilize the Phase 1 Saturn analyzer and test menu to expand the capacity beyond antiplatelet therapy (APT) assessment and monitoring to include general platelet dysfunction that is not APT-specific.

The Phase 2 analyzer will utilize an updated algorithm that can reliably conduct platelet function measurements over an expanded hematocrit range (≥21% HCT) and will have an increased menu offering.

At a minimum, data analysis will be performed using the latest version of CLSI EP09-A3 and EP12-A2 as guidelines with Analyse-it/Microsoft Excel or similar software. Additional analysis may be added as required.

The estimated sample size in this study is expected to yield results to allow continued development of the Saturn Investigational Instrument and is based on prior translational clinical experience with similar device development activities. There has been no formal power analysis, and the population size is not intended to support a regulatory submission.

The purpose of this evaluation is to gain information on the system functionality and analytical performance of the Saturn Investigational Instrument using whole blood samples. One Saturn cartridge will be tested in parallel with Chronolog LTA for each patient.

This is an observational study that will be conducted in patients undergoing open heart surgery. The outcome of this evaluation will be used to inform future development activities. Data will not be used in a regulatory submission.

Recruitment will occur at Sinai Hospital of Baltimore. The expected length of recruitment period is up to 6 months. A minimum of 75 patients are expected to participate in this trial. Patient participation will entail pre-, intra-, and peri-operative phlebotomy up to 48 hours after surgery. In-hospital clinical and outcome data will be collected. Subject consent to participate in the research will be documented by the investigator per the institution policies regarding informed consent and 21 CFR part 50.

The screening process will consist of routine preoperative screening, which is part of the standard of care prior to cardiac surgery. Preoperative medical evaluation will include review of patient's history, physical examination, and available cardiac and other diagnostic risks for the proposed operation. Those who meet all inclusion criteria and none of the exclusionary criteria are eligible for enrollment.

All patients will undergo standardized anesthesia and surgical protocol. Blood samples will be collected and analyzed at the following timepoints: pre-anesthesia, immediately post-protamine (off pump), 1-2 hours post-protamine and up to 48 hours post-surgical completion. A total of up to 60 ml (up to 15ml at each timepoint) of blood will be collected for research purposes throughout the study duration. Blood sampling will be obtained via a central venous catheter or direct phlebotomy depending on the time of CVC discontinuation. Medical records will be reviewed to assess for in-hospital serious adverse events and to document blood loss, bleeding events, and blood transfusion requirements.

All laboratory assessments will be completed prior to anesthesia induction, immediately post-protamine, 1-2 hours post-protamine and up to 48 hours post-surgical completion.

* Saturn Investigational Cartridge
* Light transmittance platelet aggregation stimulated by collagen, ADP, TRAP, and arachidonic acid
* CBC

The study is comprised of 4 periods: Preoperative and screening, during surgery, after surgical completion, and in-hospital pre-discharge. The preoperative and screening period is comprised of baseline assessments and assessment of safety laboratory values and platelet function testing. During surgery and after surgical completion assessments are comprised of safety laboratory and platelet function testing while in-hospital pre-discharge assessment is comprised mainly of adverse and bleeding events via medical records review.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age
* Subject scheduled for elective cardiothoracic surgery requiring a sternotomy
* Coronary artery bypass grafting (CABG)
* Combined CABG and valve surgery
* On-pump double or triple valve procedures
* Aortic surgery or redo surgery
* Off pump CABG as part of a hybrid revascularization approach
* Able to read and has signed and dated the informed consent form

Exclusion Criteria:

* Subject requiring an emergency procedure
* Pregnancy
* Subject is hemodynamically unstable
* Conversion to on-pump
* History of bleeding tendencies
* History of coagulation disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sinai Hospital of Baltimore
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2022-03-23 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
System functionality and analytical performance of Saturn Investigational Instrument and Cartridge | 48 hours after open heart surgery
  Comparison of platelet aggregation between Saturn Investigational Instrument and Light Transmittance Aggregation

CONTACTS AND LOCATIONS:
Overall Officials: Paul Gurbel, MD, Principal Investigator — Sinai Center for Thrombosis Research and Drug Development
Locations (1):
- Sinai Center for Thrombosis Research, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Do not plan to share IPD.